CLINICAL TRIAL: NCT01688466
Title: A Randomized Phase 2 Single-Center Study of Pomalidomide for Chronic GvHD
Brief Title: Pomalidomide for Chronic Graft-versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Najla El Jurdi, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120197; 12-C-0197
Record Dates: First submitted 2012-09-15; First posted 2012-09-20 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Graft vs Host Disease; Graft-Versus-Host Disease
Keywords: Immune Modulatory; Systemic Absorption; Oral Agent
MeSH Terms: conditions — Graft vs Host Disease | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.5 mg/day with Dose Escalation (Experimental): 0.5 mg/day with Dose Escalation by 0.5 mg/day increments every 2 weeks to a maximum of 2.0 mg/day
  Interventions: Drug: Pomalidomide
- 0.5 mg/day without Dose Escalation (Experimental): 0.5 mg/day without Dose Escalation
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — 0.5 mg/day with and/or without Dose Escalation and 0.5 mg/day- 2.0 mg/day by mouth (PO) QD(every day) of each 28 day cycle
  Other Names: POMALYST

SUMMARY:
Background:

- Pomalidomide is a drug that alters the body's immune response. It may help people who have chronic graft-versus-host disease (GvHD). GvHD may appear after a stem cell transplant, when immune cells in the transplant try to attack tissues in the person who received the transplant. GvHD is not easy to treat, and often does not respond to standard treatments. Researchers want to see if pomalidomide is a safe and effective treatment for GvHD.

Objectives:

- To test the safety and effectiveness of pomalidomide for GvHD that has not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have GvHD that has not responded to standard treatments.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will also be collected. A lung function test and imaging studies will also be given.
* Participants will take pomalidomide capsules once a day for 4-week periods called cycles.
* Treatment will be monitored with frequent blood tests and imaging studies. Saliva samples and skin and mouth tissue biopsies will also be collected during treatment.
* Treatment will continue for six cycles (6 months), unless the GvHD gets worse or side effects are too severe. If the GvHD has improved at the end of the six cycles, participants may be able to continue to take pomalidomide for up to six more cycles.

DETAILED DESCRIPTION:
BACKGROUND:

* Chronic graft-versus-host disease (cGvHD) is the leading cause of non-relapse morbidity and mortality in persons after allogeneic hematopoietic cell transplants.
* About 50% of persons with cGvHD have disease refractory to systemic corticosteroids and there is no standard second-line therapy.
* Thalidomide, a drug with immune-modulating effects, was active in advanced cGvHD but was difficult to use at appropriate doses.
* Pomalidomide is related to thalidomide but with higher potency and more favorable toxicity profile. It is active in multiple myeloma and myeloproliferative neoplasm associated myelofibrosis. Preliminary data in humans with cGvHD are encouraging but data are limited.

OBJECTIVES:

- Primary: Determine whether pomalidomide is effective in persons with moderate or severe cGvHD not controlled by corticosteroids.

ELIGIBILITY:

Inclusion Criteria

* Moderate or severe cGvHD per National Institutes of Health (NIH) criteria
* Age 18 to 75 years old
* Karnofsky performance score greater than or equal to 60%
* Has cGvHD that did not respond to high-dose corticosteroids (average 0.5 mg/kg/d prednisone for greater than or equal to 8 weeks) or second-line therapy
* Receiving stable or tapering doses of systemic therapy in the preceding 4 weeks
* Agree to adhere to methods of contraception and other fertility control measures as prescribed by the protocol

Exclusion Criteria

* Acute GvHD (classic and late per NIH criteria)
* Absolute neutrophils <1.0x10(9)/L, platelets <75x10(9)/L, estimated creatinine clearance <50 mL/min/1.73m(2)
* NIH lung score 3
* Pregnant or lactating
* Uncontrolled infection

DESIGN:

Randomized phase 2 trial with the single stage selection design. Patients will receive either a constant low dose of pomalidomide (0.5 mg/day) for six months or a strategy of increasing dose of pomalidomide from 0.5 mg/d up through each individual patient's maximum tolerated dose, with escalations by 0.5 mg/d every 2 weeks to a maximum of 2.0 mg/d. As an early stopping rule for futility, if after 7 patients have enrolled on either arm, 0 have responded, then no further patients will be accrued to that arm as soon as this can be determined. To protect patient safety, an early stopping rule will be implemented. With two arms, each of which has a maximal accrual of 16 patients, up to 32 evaluable patients will be randomized. Response assessments will occur every 3 months with primary efficacy endpoint evaluated at 6 months. Patients with responding disease will continue therapy for another 6 months.

ELIGIBILITY:
* INCLUSION CRITERIA
* Moderate or severe chronic graft-versus-host disease (cGvHD) diagnosed and staged per National Institutes of Health (NIH) criteria
* Greater than or equal to18-75 years of age, because no dosing or adverse event data are currently available on the use of pomalidomide in persons greater than or equal to18 years of age
* Has cGvHD that did not respond to high-dose corticosteroids (average 0.5 mg/kg/d prednisone for >8 weeks) or second-line systemic therapy
* If taking systemic therapy for cGvHD at the time of enrollment, must be on a stable or tapering schedule in the preceding 4 weeks (extracorporeal photopheresis has to be stopped at least by 4 weeks before enrollment)
* Karnofsky performance score greater than or equal to 60%
* Life expectancy >3 months
* Stable primary malignancy for previous 3 months
* Agree to adhere to methods of contraception and other fertility control measures as prescribed by the protocol
* Because agents of this class are known to be teratogenic, women of childbearing potential and men must agree to use effective forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Females of childbearing potential (FCBP) (Cross) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10

  14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods, AND Education and Counseling Guidance Document.
* Male Subjects
* Must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation of study drug even if he has undergone a successful vasectomy
* Will be warned that sharing study drug is prohibited and will be counseled about pregnancy precautions and potential risks of fetal exposure
* Must agree to abstain from donating blood, semen, or sperm during study participation and for at least 28 days after discontinuation of study drug.
* Must agree that if a pregnancy or a positive pregnancy test does occur in a study subject or the partner of a male study subject during study participation, study drug must be immediately discontinued.
* Patients must agree to not share study drug with anyone during participation in the study.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* All study participants must be registered into the mandatory POMALYST REMS (TM) program, and be willing and able to comply with the requirements of the POMALYST REMS (TM) program.

EXCLUSION CRITERIA:

* Acute GvHD, classic (less than or equal to day 100) or late-onset (>day 100)
* Systemic immune suppression or systemic therapy for cGvHD started within preceding 4 weeks including extracorporeal photopheresis
* Hypersensitivity to thalidomide, lenalidomide or pomalidomide
* Any serious medical condition which places the subject at an unacceptable risk if he or she were to participate in the study or confounds the ability to interpret data from the study, including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Neutrophil <1.0x10(9)/L, platelets <75x10(9)/L, estimated creatinine clearance <50 mL/min/1.73m(2) (Cockroft-Gault formula) total bilirubin >3 mg/dL, transaminase>3xUNL
* Uncontrolled infection
* Active human immunodeficiency virus 1 (HIV-1), hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection

Uncontrolled arrhythmias or symptomatic heart disease or left ventricular ejection fraction (LVEF) <45%

* Other cancer except that for which the transplant was done <2 years before study entry, except non-melanoma skin cancer or carcinoma in situ of the uterine cervix or breast
* Taking other investigational drugs
* NIH lung score 3
* Pregnant women are excluded from this study because pomalidomide has potential for teratogenic effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pomalidomide, breastfeeding must be discontinued while the mother is taking study drug and for at least 28 days after discontinuation of study drug. These potential risks may also apply to other agents used in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-08-30 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Jurdi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolanos-Meade J, Vogelsang GB. Chronic graft-versus-host disease. Curr Pharm Des. 2008;14(20):1974-86. doi: 10.2174/138161208785061373. PMID 18691108
- [Background] Lee SJ, Vogelsang G, Flowers ME. Chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2003 Apr;9(4):215-33. doi: 10.1053/bbmt.2003.50026. PMID 12720215
- [Background] Martin PJ, Weisdorf D, Przepiorka D, Hirschfeld S, Farrell A, Rizzo JD, Foley R, Socie G, Carter S, Couriel D, Schultz KR, Flowers ME, Filipovich AH, Saliba R, Vogelsang GB, Pavletic SZ, Lee SJ; Design of Clinical Trials Working Group. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: VI. Design of Clinical Trials Working Group report. Biol Blood Marrow Transplant. 2006 May;12(5):491-505. doi: 10.1016/j.bbmt.2006.03.004. PMID 16635784
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0197.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.5 mg/Day With Dose Escalation | 0.5 mg/Day Without Dose Escalation
Started | 17 | 17
Completed | 15 | 10
Not Completed | 2 | 7
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 4
Not completed — Not evaluable | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 mg/Day With Dose Escalation | 0.5 mg/Day Without Dose Escalation | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (14.2) | 46.8 (13.9) | 47.65 (14.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 10 | 12 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 15 | 17 | 32
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mexican, Puerto Rican, Cuban, Central/So. American | 0 | 2 | 2
  Not meeting definition for Hispanic or Latino | 17 | 15 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Response at 6 Months
Description: Overall response was assessed by the National Institutes of Health (NIH) Chronic Graft-Versus Host Disease (cGVHD) Response criteria. Complete response (CR) is complete resolution in all signs and symptoms at all affected organs or tissues. Partial response (PR) is improvement in ≥ 1 organ or tissue with no progression in any other affected organ or tissue. Response < PR is a change towards improvement from the pre-treatment baseline but not meeting the criteria for CR or PR. Stable disease (SD) is no change in cGVHD. Flare is exacerbation of cGVHD manifestations during withdrawal of immunosuppressive therapy which do not exceed those at the beginning of the trial and improves after reinstatement of previous treatment. Progressive disease (PD) is failure of therapy to control cGVHD . Mixed response (improvement in some organs but worsening in others) will be categorized as progressive disease.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg/Day With Dose Escalation | 0.5 mg/Day Without Dose Escalation
Number analyzed (Participants) | 17 | 17
Participants
  Complete Response | 0 | 0
  Partial Response | 7 | 9
  Progressive Disease | 2 | 5
  Stable Disease | 0 | 1
  Mixed Response | 0 | 0
  Response < Partial Response | 0 | 0
  Flare | 0 | 0
  Did not respond to treatment | 1 | 0
  Not Evaluable | 7 | 2

2. Secondary Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v4.0
Description: Here is the count of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v4.0. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 50 months and 20 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg/Day With Dose Escalation | 0.5 mg/Day Without Dose Escalation
Number analyzed (Participants) | 17 | 17
Participants | 17 | 17

ADVERSE EVENTS:
Time Frame: 50 months and 20 days
Arm/Group | 0.5 mg/Day With Dose Escalation | 0.5 mg/Day Without Dose Escalation
All-Cause Mortality (participants affected / at risk) | 0/17 | 1/17
Serious Adverse Events (participants affected / at risk) | 11/17 | 8/17
Other Adverse Events (participants affected / at risk) | 17/17 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg/Day With Dose Escalation (N=17) | 0.5 mg/Day Without Dose Escalation (N=17)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (1)
Carbon monoxide diffusing capacity decreased (Investigations) | 2 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) — Gastroenteritis
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) — CMV reactivation
Lung infection (Infections and infestations) | 2 (2) | 5 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Salivary gland infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 2 (4)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg/Day With Dose Escalation (N=17) | 0.5 mg/Day Without Dose Escalation (N=17)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (2)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 2 (2) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) — ST depression
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Dry eye (Eye disorders) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 10 (11) | 3 (3)
Flu like symptoms (General disorders) | 0 (0) | 2 (2)
Forced expiratory volume decreased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) — reflux + fullness
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (10) | 4 (5)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 0 (0) — throat tightness, dry mouth, pruritis
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) — CMV reactivation
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 4 (5) | 3 (3)
Lymphocyte count decreased (Investigations) | 10 (14) | 8 (9)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — L. plantar fascilitis
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (8) | 2 (2)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (7)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — increased plaques
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — leg wounds
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — upper extremity, neck tightness
Skin infection (Infections and infestations) | 1 (4) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 5 (5) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (14)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Updated Protocol and SAP (2025-04-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT01688466/Prot_SAP_003.pdf
  • Informed Consent Form: Updated Standard Consent (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT01688466/ICF_004.pdf